CLINICAL TRIAL: NCT02279472
Title: Optical Coherence Tomography Quantitative Analysis of Changes in Anterior Chamber After Laser Peripheral Lridotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Haomin Luo, Haomin Luo M.d., Second Xiangya Hospital of Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SecondXHCSU
Record Dates: First submitted 2014-09-30; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Primary Angle Closure Glaucoma
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- laser peripheral iridotomy (Other): Laser peripheral iridotomy (LPI) is widely regarded as the first-line intervention for either acute or chronic types of angle-closure glaucoma in early stage ,which relieves pupil block and thus flattening the iris contour and widening the drainage angle,performd by Nd.YAG LASER
  Interventions: Procedure: Laserex Tango Nd:YAG, Ellex-SuperQ Medical, Australia

INTERVENTIONS:
Procedure: Laserex Tango Nd:YAG, Ellex-SuperQ Medical, Australia — All the patients will be achieved with pilocarpine 1% for pupil constriction, laser peripheral iridotomy(LPI) is performed using the ophthalmic neodymium: yttrium aluminium garnet laser (Laserex Tango Nd:YAG, Ellex-SuperQ Medical, Australia) and an VOLK iridotomy contact lens. After LPI, patients will be given topical prednisolone acetate 0.1% for 7 days.

SUMMARY:
The purpose of this study is to analysis changes in anterior segment morphology after laser peripheral lrldotomy measured by optical coherence tomography, and to evaluate treatment effectiveness

DETAILED DESCRIPTION:
In the study ,primary angle closure(PAC) and primary angle closure glaucoma (PACG) will be recruited. Anterior segment optical coherence tomography images captured before and after laser peripheral iridotomy will be analysed to provide objective and reproducible quantification of anterior segment biometric parameters.The outcomes can provide useful information for clinical strategies in the treatment and management of pathology related to angle closure.

ELIGIBILITY:
Inclusion Criteria:

1 .The gonioscopy or UBM examination has confirmed the diagnosis of PACS or PAC 2. Intraocular pressure within 10 to 21 mmHg ，C/D≤0.6 3. Visual field is normal or only show paracentral scotoma 4. Vision or corrected visual acuity ≥0.8 5. Refractive degree no more than 200D 6. Exclude other ocular and systemic diseases

-

Exclusion Criteria:

1. Corneal macula and other corneal diseases, ocular surface disease or corneal edema
2. Iridocyclitis
3. Ocular trauma and intraocular operation history
4. No fixationFundus lesions such as diabetic retinopathy or retinal detachment
5. No fixation
6. Ocular or systemic application of cortical steroids -

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-10; Primary Completion 2014-12 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Changes in anterior chamber after LPI at 1 month | 1month

CONTACTS AND LOCATIONS:
Overall Officials: Xuanchu Duan, Ph.D, Study Director — Second Xiangya Hospital of Central South University
Locations (1):
- The Second Xiangya Hospital of Central South University,, Changsha, Hunan, China

REFERENCES:
- [Background] Memarzadeh F, Li Y, Chopra V, Varma R, Francis BA, Huang D. Anterior segment optical coherence tomography for imaging the anterior chamber after laser peripheral iridotomy. Am J Ophthalmol. 2007 May;143(5):877-9. doi: 10.1016/j.ajo.2006.11.055. Epub 2006 Dec 29. PMID 17452177
- [Background] Lee KS, Sung KR, Shon K, Sun JH, Lee JR. Longitudinal changes in anterior segment parameters after laser peripheral iridotomy assessed by anterior segment optical coherence tomography. Invest Ophthalmol Vis Sci. 2013 May 3;54(5):3166-70. doi: 10.1167/iovs.13-11630. PMID 23599331